CLINICAL TRIAL: NCT04394143
Title: Effect of AD128 on Obstructive Sleep Apnea Severity: a Randomized, Placebo-controlled, Double-blind, Cross-over Study
Brief Title: Effect of AD128 to Treat Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Raphael Heinzer (Other)
Collaborators: Apnimed (Industry)
Responsible Party: Sponsor-Investigator, Raphael Heinzer, Prof. Raphael Heinzer, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-00315
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Sleep Apnea, Obstructive
Keywords: obstructive sleep apnea; pharmacologic treatment; sleepiness; vigilance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleepiness | interventions — Mannitol

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, double-blind crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Evaluators, investigators and patients will be blinded to treatment allocation. Treatments will be prepared and conditioned by the Pharmacy Service of the University Hospital of Lausanne according to a randomisation list performed by an independent statistician. The Pharmacy service is completely independent from the Center for Investigation and Research in Sleep (CIRS). Unblinding will be performed after statistical analysis is completed by a statistician blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AD128 (Experimental): The study specific intervention includes per oral administration of two capsules of AD128, once daily, just before lights out, for 7 days.
  Interventions: Drug: AD128
- placebo (Placebo Comparator): Two placebo capsules (Mannitol) will be administered for the control intervention once daily, just before light outs, for one week.
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: AD128 — Oral administration of two capsules before sleep for 7 days.
  Arms: AD128
Drug: Mannitol — Oral administration of two capsules before sleep for 7 days.
  Other Names: Placebo
  Arms: placebo

SUMMARY:
This study evaluates the combination of two drugs (AD128), to treat obstructive sleep apnea (OSA) severity. After a baseline evaluation and during 7 days, half of the participants will randomly receive this drug combination (AD128) and the other will receive a placebo, i.e. a drug without pharmaceutical effect. Neither the participants, nor the investigators will know in which arm participants are until the end of the study. After one week of trial, an evaluation will be perform and will be follow by one week without any treatment. During the third and last week of trial, there will be a crossover of the groups, i.e. the participants of the first group who took the two drugs (AD128) during the first week will take a placebo and those who took the placebo will take the drugs combination.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years and ≤ 65 years)
* New or previous diagnosis of OSA with an AHI > 15/h on a polygraphic or polysomnographic recording (Participants already treated with continuous positive airway pressure (CPAP) or mandibular advancement device can be included but a 7-days wash-out period is required before the beginning of the protocol and CPAP usage will not be possible during the whole protocol duration),
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* History of seizures,
* History of glaucoma,
* History of benign prostatic hyperplasia, organic miction disorder or urinary retention,
* Gastrointestinal disease (e.g. stenosis, occlusion, ulcerative colitis, toxic megacolon, hiatal hernia…)
* Cardiac arrhythmia,
* History of bipolar disorder,
* Use of respiratory stimulants or depressants,
* Use of Hypnotics,
* Use of Central nervous system stimulants,
* Use of Monoamine oxidase inhibitors (MAOIs) antidepressant,
* Major depressive disorder,
* Central sleep apnea representing more than 10% of all respiratory events
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Pregnant or breast feeding female participants or participants who intend to become pregnant during the study (However, there is no contraindication to contraception),
* Other clinically significant concomitant disease states (renal failure, hepatic dysfunction, severe cardiovascular or respiratory disease, myasthenia gravis, cerebral sclerosis),
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Use or morphinic and derivatives which may influence sleep,
* Refusal to be informed in case of incidental findings.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | Day 7 and 21
  Change from baseline AHI (events/h) measured via polysomnography between the week of investigational treatment (AD128) and the week of placebo treatment.

SECONDARY OUTCOMES:
Oxygen desaturation index (ODI) | Day 7 and 21
  Change from baseline ODI (events/h) measured via polysomnography between the week of investigational treatment (AD128) and the week of placebo treatment.
Oxygen desaturation index (ODI) in REM and NREM | Day 7 and 21
  Change from baseline ODI (events/h) measured via polysomnography during rapid eye movement (REM) and non rapid eye movement (NREM) sleep between the week of investigational treatment (AD128) and the week of placebo treatment.
Hypoxic load | Day 7 and 21
  Change from baseline hypoxic load (area under the curve of 3% oxygen desaturation related to apnea-hypopnea events) measured via polysomnography between the week of investigational treatment (AD128) and the week of placebo treatment.
Hypoxic load in REM and NREM | Day 7 and 21
  Change from baseline hypoxic load (area under the curve of 3% oxygen desaturation related to apnea-hypopnea events) measured via polysomnography during rapid eye movement (REM) and non rapid eye movement (NREM) sleep between the week of investigational treatment (AD128) and the week of placebo treatment.
Arousal index | Day 7 and 21
  Change from baseline arousal index (events/h) measured via polysomnography between the week of investigational treatment (AD128) and the week of placebo treatment.
Arousal index in REM and NREM | Day 7 and 21
  Change from baseline arousal index (events/h) measured via polysomnography during rapid eye movement (REM) and non rapid eye movement (NREM) sleep between the week of investigational treatment (AD128) and the week of placebo treatment.
Pulse wave amplitude (PWA) drops | Day 7 and 21
  Change from baseline PWA drops (events/h) measured via polysomnography between the week of investigational treatment (AD128) and the week of placebo treatment.
Pulse wave amplitude (PWA) drops in REM and NREM | Day 7 and 21
  Change from baseline PWA drops (events/h) measured via polysomnography during rapid eye movement (REM) and non rapid eye movement (NREM) sleep between the week of investigational treatment (AD128) and the week of placebo treatment.
Apnea-hypopnea index (AHI) in REM and NREM | Day 7 and 21
  Change from baseline AHI (events/h) measured via polysomnography during rapid eye movement (REM) and non rapid eye movement (NREM) sleep between the week of investigational treatment (AD128) and the week of placebo treatment.
Percentage of REM sleep | Day 7 and 21
  Change from baseline REM sleep (% of total sleep time) measured via polysomnography between the week of investigational treatment (AD128) and the week of placebo treatment.
Percentage of N1 | Day 7 and 21
  Change from baseline sleep stage 1 (N1: % of total sleep time) measured via polysomnography between the week of investigational treatment (AD128) and the week of placebo treatment.
Percentage of N2 | Day 7 and 21
  Change from baseline sleep stage 2 (N2: % of total sleep time) measured via polysomnography between the week of investigational treatment (AD128) and the week of placebo treatment.
Percentage of N3 | Day 7 and 21
  Change from baseline sleep stage 3 (N3: % of total sleep time) measured via polysomnography between the week of investigational treatment (AD128) and the week of placebo treatment.
Percentage of alpha wave | Day 7 and 21
  Change from baseline alpha wave frequency (8-13 Hz - % of total sleep time) measured via polysomnography in REM and NREM between the week of investigational treatment (AD128) and the week of placebo treatment.
Percentage of beta wave | Day 7 and 21
  Change from baseline beta wave frequency (13-30 Hz - % of total sleep time) measured via polysomnography in REM and NREM between the week of investigational treatment (AD-128) and the week of placebo treatment.
Percentage of gamma wave | Day 7 and 21
  Change from baseline gamma wave frequency (30-100 Hz - % of total sleep time) measured via polysomnography in REM and NREM between the week of investigational treatment (AD128) and the week of placebo treatment.
Percentage of theta wave | Day 7 and 21
  Change from baseline theta wave frequency (4-8 Hz - % of total sleep time) measured via polysomnography in REM and NREM between the week of investigational treatment (AD128) and the week of placebo treatment.
Percentage of delta wave | Day 7 and 21
  Change from baseline delta wave frequency (1-4 Hz - % of total sleep time) measured via polysomnography in REM and NREM between the week of investigational treatment (AD128) and the week of placebo treatment.
Reaction time PVT | Day 7 and 21
  Change from baseline reaction time (in ms) during Psychomotor Vigilance Task (PVT). During 10 min, subjects were instructed to press a button as quickly as possible when a red millisecond-counter appeared on a small screen (PVT-192, Ambulatory Monitoring Inc.).
Lapse PVT | Day 7 and 21
  Change from baseline lapse time (in ms) during Psychomotor Vigilance Task (PVT) and defined as reaction time > 500 ms). During 10 min, subjects were instructed to press a button as quickly as possible when a red millisecond-counter appeared on a small screen (PVT-192, Ambulatory Monitoring Inc.).
Chronic Excessive daytime sleepiness (EDS) | Day 7 and 21
  Change from baseline Epworth Sleepiness Scale (ESS) score between the week of investigational treatment (AD128) and the week of placebo treatment.
  The ESS is a 8-item questionnaire. ESS score can range from 0 to 24. The higher the ESS score, the higher daytime sleepiness.
Acute Excessive daytime sleepiness (EDS) | Day 7 and 21
  Change from baseline Stanford Sleepiness Scale (SSS) score between the week of investigational treatment (AD128) and the week of placebo treatment.
  Consisting of only one item, the scale requires respondents to select one of seven statements best representing their level of perceived sleepiness. The scale range from 1 to 7. Higher score indicates greater sleepiness.
Sleep quality | Day 7 and 21
  Change from baseline visual analogic scale (VAS) sleep quality score between the week of investigational treatment (AD128) and the week of placebo treatment. Score ranges from 0 to 10. Higher score indicates better sleep quality.
Fatigue | Day 7 and 21
  Change from baseline Pichot scale score between the week of investigational treatment (AD128) and the week of placebo treatment.
  The Pichot scale is a 8-items auto-questionnaire to assess excessive fatigue. Score varies between 0 and 32, a score > 22 indicates excessive fatigue.
Systolic and diastolic blood pressure | Day 7 and 21
  Change from baseline office systolic and diastolic blood pressure (BP in mm Hg) between the week of investigational treatment (AD128) and the week of placebo treatment.
  The Pichot scale is a 8-items auto-questionnaire to assess excessive fatigue. Score varies between 0 and 32, a score > 22 indicates excessive fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Heinzer, MD, Principal Investigator — University Hospital of Lausanne (CHUV)
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) could be transmitted on request after publication to researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Berger M, Solelhac G, Marchi NA, Dussez R, Bradley B, Lecciso G, Heiniger G, Bayon V, Van Den Broecke S, Haba-Rubio J, Siclari F, Heinzer R. Effect of oxybutynin and reboxetine on obstructive sleep apnea: a randomized, placebo-controlled, double-blind, crossover trial. Sleep. 2023 Jul 11;46(7):zsad051. doi: 10.1093/sleep/zsad051. PMID 36861433